CLINICAL TRIAL: NCT05794399
Title: Comparison of Warfarin Versus Rivaroxaban in Management of Post-myocardial Infarction Left Ventricular Thrombus in a Tertiary Cardiac Center of Nepal: a Randomized Control Study.
Brief Title: Anticoagulation in Post MI LV Thrombus Trial in Nepal
Acronym: WaRMIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Gangalal National Heart Centre (Other)
Responsible Party: Principal Investigator, Dipanker Prajapati, Consultant Cardiologist, Shahid Gangalal National Heart Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGNHC-RCT
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Left Ventricular Thrombus; Myocardial Infarction
Keywords: Post Myocardial Infarction; Left Ventricular Thrombus; Warfarin; Rivaroxaban; Nepal
MeSH Terms: conditions — Myocardial Infarction | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: 1:1 parallel study design
Who Masked: Outcomes Assessor
Masking Description: The radiologist who will assess the presence or absence of left ventricular (LV) thrombus will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): In this arm, the patients with post-myocardial infarction and left ventricular thrombus will be treated with Rivaroxaban 20mg or 15mg as indicated.
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): In this arm, the patients with post-myocardial infarction and left ventricular thrombus will be treated with warfarin with a dose adjusted with the International Normalised ratio range of 2.0 to 3.0.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Intervention Group:
  The patients in the intervention group will be treated with Rivaroxaban 20 mg once daily with the evening meal in patients with a CrCl >50 mL/min OR 15 mg in cases of moderate-to-severe renal impairment dose with the dosing of once daily with the evening meal in patients with a CrCl ≤50 mL/min. The patient in the intervention group will be requested for follow-up after 3 months of commencing the treatment or whenever the signs and symptoms of bleeding events are noted.
  Arms: Rivaroxaban
Drug: Warfarin — Control Group:
  The patients in the control group will be treated with Warfarin. The dose will be started with 5 mg and will be titrated based on the International Normalized Ratio (INR) which will be targeted at the range of 2.0 to 3.0. The dual antiplatelet duration will be based on the latest guidelines. The patients will be asked for frequent INR monitoring on an OPD basis until the INR is within the therapeutic range, after which patients will be asked for monthly follow-up INR reports. The patients in the control group will not be treated with heparin or low molecular weight heparin before the INR is maintained in the therapeutic range.
  Arms: Warfarin

SUMMARY:
Introduction:

The prevalence of left ventricular(LV) thrombus after acute myocardial infarction has decreased with thrombolysis and primary angioplasty intervention worldwide. However, most of the patients in our country present late after the onset of ischemia resulting in a comparable increase proportion of late presentation MI compared to developed countries. This delayed presentation is associated with the increased incidence of LV thrombus, associated with increased cerebrovascular and cardiovascular events resulting in increased morbidity and mortality. The Vitamin K Antagonist Warfarin is indicated in recent guidelines for the duration of 3-6 months. The use of Warfarin is less in our part of the world due to the requirement of frequent International Normalized Ration (INR) monitoring and dietary restrictions. Novel oral anticoagulants (NOACs) are an alternate option for such hindrance to the treatment of LV thrombus. This research will help assess the safety and efficacy of Rivaroxaban, one of the NOACs compared to warfarin.

Objectives:

Our aim will be to compare the efficacy of rivaroxaban compared to warfarin in the complete resolution of post-MI LV thrombus. The primary efficacy endpoint of our study will be a resolution of LV thrombus as assessed by cardiac MRI at the end of 3 months of the study period. The secondary endpoint will be the comparison of the safety of both drugs measured by the incidence of major bleeding and embolic events.

Methods:

The patients who present late after acute MI in our center with LV thrombus will be enrolled in our study. The diagnosis of LV thrombus will be diagnosed by cardiac MRI, which is considered the gold standard for the diagnosis. The patients then will be randomized in a 1:1 ratio to either warfarin or rivaroxaban within 24 hours of diagnosis of LV thrombus. The warfarin group will be prescribed the warfarin in the dose of 5mg daily and the dose titrated according to the INR value to maintain the INR range of 2 to 3. Rivaroxaban group will be prescribed 15 to 20mg according to the indication. The research group consisting of the principal investigator and coinvestigators will be responsible for the recruitment and overall study procedures.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality and morbidity among non-communicable diseases worldwide including in Nepal. Myocardial infarction(MI) is the main disease among cardiovascular diseases. [i] MI is also the main reason for hospitalization in the cardiac centers of our country. [ii] There is an additional burden of late presentation of MI in our setting due to lack of proper awareness, limited access to health care and improper referral mechanism. In the hospital-based registry in 2018, more than 65% of acute MI presented after the eligible time frame for primary angioplasty or thrombolysis. [iii] The incidence of the formation of left ventricular (LV) thrombus is increased with the late presentation. Worldwide, the prevalence of LV thrombus before the era of primary angioplasty was around 31-57%. [iv],[v],[vi] After the start of the primary angioplasty techniques, the prevalence of post-MI LV thrombus has decreased to around 15%.[vii] However, it is still associated with increased risks of embolic events and mortality.[viii],[ix],[x] European and American guidelines have recommended using vitamin K antagonist (VKA) for a minimum of 3-6 months as a class IIa, LOE c, with duration individualized to bleeding risk with a target of international normalized ratio (INR) of 2.5 (range of 2 to 3). [xi],[xii] Non-VKA oral anticoagulants (NOACs) in addition to the dual antiplatelet therapy in these patients are attractive alternatives because of their potential efficacy and safety along with ease of administration, lack of requirement for INR monitoring or dietary restrictions resulting in overall improvement of life.[xiii] However, there is no randomized control trial comparing warfarin and NOACs. There are two ongoing trials NCT01556659 and NCT03764241. The recommendation is more relevant to us as there is an overburden of patients presenting late due to various geographical and financial reasons. This study was designed for the evaluation of anticoagulation effects among the acute ST elevation Myocardial Infarction (STEMI) with LV thrombus in complete resolution of LV thrombus. The investigators aim to compare Warfarin to Rivaroxaban in the management of post-myocardial infarction left ventricular thrombus in our part of the world.

Data management and Analysis Plan:

Independent data safety and monitoring board will be formed and will be responsible for the safety concerns of the research participants. Data will be collected and entered in the computer-based CRF constructed using the password-protected free software at https://www.kobotoolbox.org. The data will be accessed by the principal investigator and the research officer only. The data will be anonymized before statistical analysis which will be performed by the separate coinvestigators responsible for the data analysis. Appropriate statistical tests will be used for measuring association and correlation. A 'P' value of less than 0.05 will be considered to be significant.

Dissemination Plan:

The findings of the study will be published in a peer-reviewed journal and presented at national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years hospitalized with the diagnosis of acute STEMI and
* Presence of LV thrombus which is confirmed with cardiac MRI.

Exclusion Criteria:

1. Bleeding risk Active bleeding; history of intracranial hemorrhage; clinically significant gastrointestinal bleeding within 12 months before randomization; severe thrombocytopenia (<50×109/L), or anemia (i.e., hemoglobin <90 g/L) at screening or pre-randomization; Liver function Child-Pugh B or C; untreated arterial aneurysm, arterial or venous malformation and aorta dissection; and body weight <40 kg.
2. Undergoing anticoagulation therapy
3. Cardiovascular condition Cardiac shock; uncontrolled blood pressure (SBP ≥180 mmHg); planned CABG within 3 months; suspicious Pseudo-ventricular aneurysm
4. Concomitant diseases Severe chronic or acute renal failure (CrCl <50 mL/min at screening or pre-randomization); significant liver disease; current substance abuse (drug or alcohol) problem; life expectancy to less than 12 months; Known allergies, or intolerance to rivaroxaban; Woman who is currently pregnant, or breastfeeding; and Other hypercoagulable states, such as a malignant tumor, SLE
5. Other conditions adjudicated by investigators to be unsuitable for anticoagulation
6. Pregnant women and participants with any cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
LV thrombus resolution | 3 months
  The primary endpoint will be a resolution of LV thrombus as assessed by cardiac MRI in 3 months of study.

SECONDARY OUTCOMES:
Major bleeding events | 3 months
  The major bleeding events will be defined according to the definition of major bleeding for non-surgical patients according to the International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC)[xiv] which is
  1. Fatal bleeding. and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or
  3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Embolic events | 3 months
  Embolic events will be defined as Cardioembolic stroke that is stroke attributable to arterial occlusion from an embolus that presumably arose in the heart. Ischemic stroke in the vascular distribution of a major intracranial or extracranial artery with >50% stenosis or occlusion on vascular imaging. Clinical findings include those of cerebral cortical involvement or brainstem or cerebellar dysfunction. Cortical and cerebellar lesions and brainstem or subcortical lesions >1.5 cm are considered potentially caused by large artery atherosclerosis. Evidence of a previous TIA or stroke in >1 vascular territory supports a clinical diagnosis of cardioembolic stroke.[xv]

CONTACTS AND LOCATIONS:
Locations (1):
- Nepal Health Research Council, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
The data safety and monitoring board will be formed which will be responsible for safety supervision and monitoring among our study participants. The board will include three members each from the Department of Cardiology, the Department of Cardiac Surgery and the Department of Cardiac Anesthesia. The board will be responsible for the safety of the study participants. The principal investigator will be primarily responsible for the entire research. A well-trained research officer will be hired who will be responsible for the recruitment of the participants, obtaining consent forms and informing the principal investigator regarding the allocation of the treatment group. The principal investigator along with the coinvestigators will be primarily responsible for the treatment of the patients and drug dosage escalation/de-escalation according to the INR report. The quality of the data will be ensured by regular data monitoring by the principal investigator.

REFERENCES:
- [Background] Bhattarai S, Aryal A, Pyakurel M, Bajracharya S, Baral P, Citrin D, Cox H, Dhimal M, Fitzpatrick A, Jha AK, Jha N, Karmacharya BM, Koju R, Maharjan R, Oli N, Pyakurel P, Sapkota BP, Shrestha R, Shrestha S, Spiegelman D, Vaidya A, Shrestha A. Cardiovascular disease trends in Nepal - An analysis of global burden of disease data 2017. Int J Cardiol Heart Vasc. 2020 Jul 31;30:100602. doi: 10.1016/j.ijcha.2020.100602. eCollection 2020 Oct. PMID 32775605
- [Background] Adhikari, C. M., Acharya, K. P., Manandhar, R., Sherpa, K., Tamrakar, R., Bogati, A., Singh, S. K., Kansakar, S., Yadav, D. N., Dhungana, M., Dhungel, S., Baniya, B., Joshi, S., Rajbhandari, S., Pandey, R., Raut, R., Prajapati, D., KC, S. S., Adhikari, J., Adhikari, A., Gautam, B., Najmy, S., Poudel, R., Timalsina, B. K., Karki, P., Poudel, S., Thakur, K. K., Limbu, D., Nepal, H. P., Sharma, M., Rauniyar, B. K., Rajbhandari, R., Limbu, Y. R., Maskey, A., Malla, R., Sharma, D., & KC, M. B. (2020). Shahid Gangalal National Heart Centre-ST-elevation Myocardial infarction Registry (SGNHC-STEMI-Registry), Nepal. Nepalese Heart Journal, 17(1), 7-16. https://doi.org/10.3126/njh.v17i1.28795
- [Background] Gottdiener JS, Gay JA, VanVoorhees L, DiBianco R, Fletcher RD. Frequency and embolic potential of left ventricular thrombus in dilated cardiomyopathy: assessment by 2-dimensional echocardiography. Am J Cardiol. 1983 Dec 1;52(10):1281-5. doi: 10.1016/0002-9149(83)90588-x. PMID 6650417
- [Background] Gottdiener JS, Massie B, Ammons SB, et al. Prevalence of left ventricular thrombus in dilated cardiomyopathy: the WATCH trial. J Am J Cardiol 2003;41:202.
- [Background] Srichai MB, Junor C, Rodriguez LL, Stillman AE, Grimm RA, Lieber ML, Weaver JA, Smedira NG, White RD. Clinical, imaging, and pathological characteristics of left ventricular thrombus: a comparison of contrast-enhanced magnetic resonance imaging, transthoracic echocardiography, and transesophageal echocardiography with surgical or pathological validation. Am Heart J. 2006 Jul;152(1):75-84. doi: 10.1016/j.ahj.2005.08.021. PMID 16824834
- [Background] Keeley EC, Hillis LD. Left ventricular mural thrombus after acute myocardial infarction. Clin Cardiol. 1996 Feb;19(2):83-6. doi: 10.1002/clc.4960190203. PMID 8821415
- [Background] Pizzetti G, Belotti G, Margonato A, Carlino M, Gerosa S, Carandente O, Chierchia SL. Thrombolytic therapy reduces the incidence of left ventricular thrombus after anterior myocardial infarction. Relationship to vessel patency and infarct size. Eur Heart J. 1996 Mar;17(3):421-8. doi: 10.1093/oxfordjournals.eurheartj.a014875. PMID 8737217
- [Background] Bhatnagar SK, al-Yusuf AR. Effects of intravenous recombinant tissue-type plasminogen activator therapy on the incidence and associations of left ventricular thrombus in patients with a first acute Q wave anterior myocardial infarction. Am Heart J. 1991 Nov;122(5):1251-6. doi: 10.1016/0002-8703(91)90563-w. PMID 1659166
- [Background] Ezekowitz MD, Wilson DA, Smith EO, Burow RD, Harrison LH Jr, Parker DE, Elkins RC, Peyton M, Taylor FB. Comparison of Indium-111 platelet scintigraphy and two-dimensional echocardiography in the diagnosis of left ventricular thrombi. N Engl J Med. 1982 Jun 24;306(25):1509-13. doi: 10.1056/NEJM198206243062502. PMID 7078607
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Keita I, Aubin-Auger I, Lalanne C, Aubert JP, Chassany O, Duracinsky M, Mahe I. Assessment of quality of life, satisfaction with anticoagulation therapy, and adherence to treatment in patients receiving long-course vitamin K antagonists or direct oral anticoagulants for venous thromboembolism. Patient Prefer Adherence. 2017 Sep 25;11:1625-1634. doi: 10.2147/PPA.S131157. eCollection 2017. PMID 29026288
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Saleh Y, Al-Abcha A, Abdelkarim O, Elwany M, Abdelfattah OM, Abdelnabi M, Almaghraby A. Meta-Analysis Comparing the Effect of Rivaroxaban Versus Vitamin K Antagonists for Treatment of Left Ventricular Thrombi. Am J Cardiol. 2021 Dec 15;161:123-125. doi: 10.1016/j.amjcard.2021.09.009. Epub 2021 Oct 14. No abstract available. PMID 34656296